CLINICAL TRIAL: NCT01883544
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, Multiple IV Administration, Sequential-Cohort, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ALXN1007 in Healthy Male and Female Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ALXN1007 in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALXN1007-US-HV-102
Record Dates: First submitted 2013-06-19; First posted 2013-06-21 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Subjects
Keywords: Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; ALXN1007; Healthy Male and Female Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALXN1007 (Experimental): Infusion of ALXN1007
  Interventions: Drug: ALXN1007
- placebo (Placebo Comparator): Infusion placebo
  Interventions: Drug: ALXN1007

INTERVENTIONS:
Drug: ALXN1007

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple intravenous (IV) doses of ALXN1007 in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy male or female (not of childbearing potential) subjects ≥25 and ≤55 years old.

2. QTcF ≤450 msec and ≤470 for females. 3. Willing and able to give written informed consent and comply with the study visit schedule.

4. Male subject and his female spouse/partner who is of childbearing potential must be using highly effective congraception1 consisting of two forms of birth control (at least one of which must be a barrier method) starting at Screening and continuing until the end of study.

1. Highly effective contraception is defined as:

   * Established use of oral, injected or implanted hormonal methods of contraception.
   * Placement of an intrauterine device or intrauterine system.
   * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.

     5. Male subjects must not donate sperm starting at Screening until the end of study.

     6. Documented vaccination with meningococcal conjugate vaccine (MCV4) at least 14 days and not more than 5 years, prior to dosing.

Exclusion Criteria:

Female subjects of childbearing potential, including any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Postmenopausal is defined as:

* Amenorrhea ≥ 12 consecutive months without another cause and a documented serum follicle stimulating hormone (FSH) level >35 mIU/mL or
* Female subjects with irregular menstrual periods and a documented serum FSH level > 35 mIU/mL.
* Women on hormone replacement therapy (HRT). Women who are using oral contraceptives, other hormonal contraceptives (i.e., vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (i.e., diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential.

  2. Positive serum pregnancy test at Screening or Day -1. 3. Serum creatinine great than the upper limit of normal (ULN) of the testing laboratory at Screening and Day -1.

  4. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >ULN of the testing laboratory at Screening and Day -1.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of multiple, IV doses of ALXN1007 in healthy male and female subjects as assessed by physical exam, vital signs, electrocardiogram (ECG), immunogenicity, laboratory analysis, and assessment of adverse events (AEs | 90 days follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- PAREXEL Baltimore EPCU, Baltimore, Maryland, United States